CLINICAL TRIAL: NCT06487195
Title: Effectiveness of a Peer-facilitated, Recovery-focused Self-illness Management Program (Peer-RESIM) for First-episode Psychosis
Brief Title: Effects of a Peer-facilitated, Recovery-focused Self-illness Management Program for First-episode Psychosis
Acronym: Peer-RESIM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Integrated Community Centers for Mental Wellness (Unknown)
Responsible Party: Principal Investigator, Prof. Wai Tong CHIEN, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 16404722
Record Dates: First submitted 2024-06-25; First posted 2024-07-05 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Psychotic Disorders
Keywords: First-episode psychosis; randomized controlled trial; peer facilitator; recovery; illness self-management; functioning
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Parallel assignment; repeated-measures, multi-centre 3-arm RCT
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Outcome assessors, researchers and clinical staff are blind to the group and intervention assignment; they are also concealed to the participant lists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Peer-facilitated, Recovery-based Self-illness-management programme (Peer-RESIM) (Experimental): The Peer-RESIM consists of 10 1.5-hour sessions (7-12 day intervals; 4 months), based on the modified CORE program manual and psychoeducation programs developed by the research team. The printed/online program is based on a self-care, personal plan for recovery workbook with 4 key components: personal recovery goals, plans to re-establish community functioning and support networks following a crisis, identifying early warning signs and creating a relapse prevention plan, and strategies and coping resources for problem-solving and maintaining wellbeing. After completing the recovery plan, participants will be empowered and supported by a peer-support worker and group members during scheduled sharing sessions.
  Interventions: Behavioral: Peer-facilitated, Recovery-based Self-illness-management programme; Behavioral: Treatment-as-usual only
- Psycho-education group (Active Comparator): The psychoeducation group (6 subgroups; 10-12 participants per group) will be led by one experienced psychiatric nurse trained in psychiatric rehabilitation and psychoeducation group programs. The program will be guided by a validated treatment protocol based on psychoeducation programs for psychotic disorders developed by the research team and McFarlane et al. The psychoeducation program consists of ten 2-hour sessions held weekly/biweekly (similar to the Peer-RESIM, completed within 4 months), with 4 key components, including introduction and goal setting; an education workshop on psychosis, treatments, and community services; group exercises and rehearsals and discussions on illness management, coping and self-care; and a summary, evaluation and future plan.
  Interventions: Behavioral: Psycho-education group; Behavioral: Treatment-as-usual only
- Treatment-as-usual only (TAU) (Other): Participants in the usual care only group (and the two intervention groups) will receive routine community mental healthcare services.
  Interventions: Behavioral: Treatment-as-usual only

INTERVENTIONS:
Behavioral: Peer-facilitated, Recovery-based Self-illness-management programme — The Peer-RESIM program will consist of 10 1.5-hour sessions (7-12 day intervals; 4 months), based on the modified CORE program workbook/manual and psychoeducation programmes developed by the research team.
  Other Names: Peer-RESIM
  Arms: Peer-facilitated, Recovery-based Self-illness-management programme (Peer-RESIM)
Behavioral: Psycho-education group — The psychoeducation group (6 subgroups; 10-12 participants per subgroup) will be led by one experienced psychiatric nurse trained in psychiatric rehabilitation and psychoeducation group programmes.
  Arms: Psycho-education group
Behavioral: Treatment-as-usual only — Participants in the TAU group will receive routine community mental healthcare services.
  Other Names: TAU

SUMMARY:
Psychosis is a major disabling and disruptive mental illness characterized by a wide variety of disturbances in cognition and emotions, resulting in poor psychosocial functioning and frequent relapses. Despite convincing evidence of short-term symptom control and functional recovery, there has been a limited amount of data generated over the past two decades on the long-term outcomes of early interventions for psychotic patients (especially, first-episode psychosis, FEP). We propose a controlled trial with an adequate study power to examine the longer-term effects (18 months) of a Peer-facilitated, Recovery-focused Self-Illness-Management program (Peer-RESIM) for adults with FEP. Specifically, the proposed study will assess the effects of better-prepared PSWs, and a culturally adapted intervention protocol designed by our multidisciplinary research team, on improving patients' self-care and recovery.

DETAILED DESCRIPTION:
People with first-episode psychosis (FEP) are often anxious/stressed and unprepared to manage the illness and associated disturbances of daily living and functioning. Due to this unpreparedness for illness management and diverse adverse health effects in FEP, different approaches to psychosocial interventions provide significant benefits in improving patients' symptom management and preventing relapses. However, similar to early interventions, inconsistent/inconclusive results have been reported for most psychosocial health outcomes, particularly over a long-term follow-up.

There is increasing evidence showing that recovery-focused care is an effective approach to community-based psychiatric rehabilitation and mental health practice. Using this approach, empowered self-help and hope cultivation can help patients develop a sense of purpose and meaning in life and optimism for the future. Peer support can be provided by ex-/co-patients with similar illness experience who have been trained to provide voluntary/in-job mental health services. Consequently, they are well-placed to model and encourage active and autonomous recovery in their peers (fellow-patients). This innovative method of supporting recovery-focused mental healthcare is increasingly popular among those developing mental healthcare services and policies.[9] However, there few high-quality trials have assessed this strategy, and there is little evidence of its positive effects on functional and clinical recovery, symptoms and hospitalizations and service satisfaction, especially in Asian countries. Structured self-help (and/or peer-supported) training and practices may have the advantage of empowering and facilitating FEP patients to meet their (co-patients') real-life personal and illness care goals; they also minimize professional input, which may enhance the feasibility, accessibility, and/or user-friendliness of an intervention and keep its cost of delivery low.

Milton and our (1st-)Co-I conducted a multi-center randomized controlled trial of peer-facilitated recovery from severe mental illness intervention in England, using the Crisis- Resolution-Team Optimisation and RElapse Prevention(CORE) program. In their trial, significantly fewer participants in the treatment group (n=120) were admitted to inpatient care (29%vs.38%), time-to-readmission was longer (112vs.86 days), and service satisfaction was higher (78%vs.41%) than the usual care only group, over a 1-year follow-up period. A similar service is required in Hong Kong, and this peer-facilitated, self-management model/approach can be adopted/tested.

Mental healthcare should maximize the self-management of individual first-episode psychosis patients' mental wellbeing, peer support, and experience-sharing for patients to improve their illness self-care and recovery. Based on the findings of Milton's and our Co-I's randomized trial of CORE program, a similar peer-facilitated, recovery-based self-illness-management program can be adopted/tested in Hong Kong, with cultural adaptations to match local service development strategies/needs.

This proposed randomized controlled trial tests two main hypotheses that:

(1) the Peer-facilitated, Recovery-focused Self-Illness-Management program (Peer-RESIM) will yield significantly greater improvements than psychoeducation and/or routine-care only at 1-week, 9-month and/or 18-month follow-ups in patients' recovery and functioning (primary outcomes).

2. It also tests the hypothesis that the Peer-RESIM will yield significantly greater improvements than the other two groups at 1-week, 9-month and/or 18-month follow-ups in psychotic symptoms, problem-solving, re-hospitalization rates, and/or service satisfaction (secondary outcomes).

The trial examines whether the Peer-RESIM participants will indicate clinically significant changes/benefits in two primary outcomes at 1-week, 9-month and/or 18-month follow-ups.

In addition, focus-group interviews will be conducted to explore the perceived benefits, service satisfaction and strengths/limitations of the Peer-RESIM from peer-facilitators' and participants' perspectives.

Methods: A assessor-blinded, three-arm multi-centre RCT was conducted. A list of 198 Chinese adult patients with FEP randomly selected from four Community Centers for Mental Wellness in Hong Kong (in 2023) (i.e., 16-17 subjects/group from each center; a total of 66 participants per group) and randomly assigned into one of the three study groups (Peer-RESIM, psycho-education, or usual care only group) by matching with computerized random numbers.

After four-month interventions, the patient outcomes will be measured at immediately, 9 months, and 18 months post-intervention, and analysed on intention-to-treat basis. Clinical significant changes in the primary outcomes will be assessed within and between groups according to Jacobson and Traux's criteria to examine the clinical benefits to patients. Focus-group interviews will also be conducted to explore the perceived benefits, service satisfaction and strengths/limitations of the Peer-RESIM from peer-facilitators' and participants' perspectives.

Study outcomes and variables:

Socio-demographic and clinical data (e.g., gender, age, clinical diagnosis, illness duration, and medications) will be collected at baseline, and changes in medications will be recorded during the study.

Primary outcomes include: the Questionnaire about the Process of Recovery (QPR) and the 43-item Specific Level of Functioning Scale.

Secondary outcomes include: the 30-item Positive and Negative Syndrome Scale (PANSS); the Revised Social-Problem-Solving Inventory (C-SPSI-R:S); Frequency and length of time to rehospitalization(s); and the 8-item Client Satisfaction Questionnaire (CSQ-8). (Note: illness/treatment insight and drug attitude as appropriate).

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese residents, aged 18-60;
* clinically and primarily diagnosed with a first-episode psychosis according to the DSM-V criteria (American Psychiatric Association 2013), and within 3 years onset of illness;
* able to understand Cantonese/Mandarin; and
* having Global Assessment of Functioning scores ≥51, indicating mild-to-moderate symptoms and challenges in maintaining work/school/family roles, but mentally stable and comprehendible to the training and education offered

Exclusion Criteria:

* recently received/are currently receiving another psychosocial or psychoeducation intervention;
* having a comorbidity of learning/cognitive/personality disorder, and/or clinically significant medical disease; or
* having a visual/language/communication difficulty/disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaire about the Process of Recovery (QPR) | Total score self-reported at recruitment
  Level of recovery from illness will be measured with the Questionnaire about the Process of Recovery (QPR) developed by Neil et al. (2009). It consists of 22 items and three subscales (self-empowerment, 10 items; effective interpersonal relationships, 6 items; and rebuilding life, 6 items). Items will be rated on a 5-point Likert scale (0, "disagree strongly" to 4, "agree strongly"; total score range, 0-88).
Questionnaire about the Process of Recovery (QPR) | Total score self-reported at 1 week post-intervention
  Level of recovery from illness will be measured with the Questionnaire about the Process of Recovery (QPR) developed by Neil et al. (2009). It consists of 22 items and three subscales (self-empowerment, 10 items; effective interpersonal relationships, 6 items; and rebuilding life, 6 items). Items will be rated on a 5-point Likert scale (0, "disagree strongly" to 4, "agree strongly"; total score range, 0-88).
Questionnaire about the Process of Recovery (QPR) | Total score self-reported at 9 months post-intervention
  Level of recovery from illness will be measured with the Questionnaire about the Process of Recovery (QPR) developed by Neil et al. (2009). It consists of 22 items and three subscales (self-empowerment, 10 items; effective interpersonal relationships, 6 items; and rebuilding life, 6 items). Items will be rated on a 5-point Likert scale (0, "disagree strongly" to 4, "agree strongly"; total score range, 0-88).
Questionnaire about the Process of Recovery (QPR) | Total score self-reported at 18 months post-intervention
  Level of recovery from illness will be measured with the Questionnaire about the Process of Recovery (QPR) developed by Neil et al. (2009). It consists of 22 items and three subscales (self-empowerment, 10 items; effective interpersonal relationships, 6 items; and rebuilding life, 6 items). Items will be rated on a 5-point Likert scale (0, "disagree strongly" to 4, "agree strongly"; total score range, 0-88).
Specific Level of Functioning Scale (SLOF) | Total score self-reported at recruitment
  Patient functioning will be measured with the 43-item Specific Level of Functioning Scale by Schneider and Struening (1983), consisting of 4 domains:- self-maintenance (12 items), social functioning (14 items), activities (11 items), and community-living skills (6 items), assessed using a 5-point Likert scale (1-"highly dependent/typical/always' to 5-"fully self-sufficient/ typical/never").
Specific Level of Functioning Scale (SLOF) | Total score self-reported at 1 week post-intervention
  Patient functioning will be measured with the 43-item Specific Level of Functioning Scale by Schneider and Struening (1983), consisting of 4 domains:- self-maintenance (12 items), social functioning (14 items), activities (11 items), and community-living skills (6 items), assessed using a 5-point Likert scale (1-"highly dependent/typical/always' to 5-"fully self-sufficient/ typical/never").
Specific Level of Functioning Scale (SLOF) | Total score self-reported at 9 months post-intervention
  Patient functioning will be measured with the 43-item Specific Level of Functioning Scale by Schneider and Struening (1983), consisting of 4 domains:- self-maintenance (12 items), social functioning (14 items), activities (11 items), and community-living skills (6 items), assessed using a 5-point Likert scale (1-"highly dependent/typical/always' to 5-"fully self-sufficient/ typical/never").
Specific Level of Functioning Scale (SLOF) | Total score self-reported at 18 months post-intervention
  Patient functioning will be measured with the 43-item Specific Level of Functioning Scale by Schneider and Struening (1983), consisting of 4 domains:- self-maintenance (12 items), social functioning (14 items), activities (11 items), and community-living skills (6 items), assessed using a 5-point Likert scale (1-"highly dependent/typical/always' to 5-"fully self-sufficient/ typical/never").

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | Changes in mean scores from recruitment to 18 months follow-up
  The 30-item Positive and Negative Syndrome Scale (PANSS) developed by Kay et al. (1987) will evaluate on three subscales: positive symptoms, negative symptoms and general psychopathology. Items will be rated on an 8-point scale (0-"absent" to 7-"extreme").
Chinese version of the Revised Social-Problem-Solving Inventory (C-SPSI-R:S) | Changes in mean scores from recruitment to 18 months follow-up
  The 25-item C-SPSI-R:S comprises two domains: problem-solving style (rational/impulsive; careless/avoidance) and orientation (positive/negative), being rated on a 5-point Likert-scale (0-"not-at-all true" to 4-"extremely true").
RE-hospitalisation rates | Changes in average rates from recruitment to 18 months follow-up
  Occurrence and time to hospitalisation, and frequency of re-hospitalisations over the past 5-6 months
8-item Client Satisfaction Questionnaire (CSQ-8) | Changes in mean scores from recruitment to 18 months follow-up
  The 8-item CSQ-8 developed by Attkisson and Zwick (1982) is a well-accepted questionnaire used to evaluate service users' opinions/comments about services received. Items are rated on a 4-point Likert scale (1-"very dissatisfied" to 4-"very satisfied").

OTHER OUTCOMES:
Perception and insight/attitude towards illness/treatment | Changes in mean scores from recruitment to 18 months follow-up
  perception and insight/attitude towards the illness and treatment, as appropriate, using valid questionnaires or qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Wai Tong Chien, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Integrated Community Centers for Mental Wellness, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
the name and email of the researchers can be shared openly for communication and collaboration.

REFERENCES:
- [Background] Chien WT, Bressington D. A randomized controlled clinical trial of a nurse-led structured psychosocial intervention program for people with first-onset mental illness in psychiatric outpatient clinics. Psychiatry Res. 2015 Sep 30;229(1-2):277-86. doi: 10.1016/j.psychres.2015.07.012. Epub 2015 Jul 10. PMID 26193827
- [Background] Johnson S, Lamb D, Marston L, Osborn D, Mason O, Henderson C, Ambler G, Milton A, Davidson M, Christoforou M, Sullivan S, Hunter R, Hindle D, Paterson B, Leverton M, Piotrowski J, Forsyth R, Mosse L, Goater N, Kelly K, Lean M, Pilling S, Morant N, Lloyd-Evans B. Peer-supported self-management for people discharged from a mental health crisis team: a randomised controlled trial. Lancet. 2018 Aug 4;392(10145):409-418. doi: 10.1016/S0140-6736(18)31470-3. PMID 30102174
- [Background] Craig TK, Garety P, Power P, Rahaman N, Colbert S, Fornells-Ambrojo M, Dunn G. The Lambeth Early Onset (LEO) Team: randomised controlled trial of the effectiveness of specialised care for early psychosis. BMJ. 2004 Nov 6;329(7474):1067. doi: 10.1136/bmj.38246.594873.7C. Epub 2004 Oct 14. PMID 15485934
- [Background] D'Zurilla TJ, Nezu A,M. Problem-solving therapy : a positive approach to clinical intervention,3rd ed. New York, NY: Springer; 2007.